CLINICAL TRIAL: NCT01394055
Title: Official Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Dose, 2-Period Crossover Study to Evaluate the Pharmacodynamics of RM-131 Administered to Patients With Diabetic Gastroparesis
Brief Title: Study to Assess Pharmacodynamics of RM-131 in Patients With Diabetic Gastroparesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RM-131-003
Record Dates: First submitted 2011-07-08; First posted 2011-07-14 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus Type 1 and 2; Diabetes Mellitus Complications; Gastroparesis; Gastrointestinal Motility Disorder
Keywords: Diabetes Mellitus Type 1 and 2; Delayed Gastric Emptying; Gastroparesis; Gastrointestinal Motility Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications; Gastroparesis | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RM-131 (Active Comparator)
  Interventions: Drug: RM-131
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-131 — 100 μg subcutaneously once
  Arms: RM-131
Drug: Placebo — Matching placebo volume subcutaneously once
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamic (PD) and pharmacokinetic (PK) profile and the safety and tolerability of RM-131 in patients with diabetes mellitus and delayed gastric emptying.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to provide written informed consent prior to any study procedures.
* Diagnosis of Type 1 or 2 diabetic gastroparesis.
* Controlled Type 1 or 2 diabetes mellitus (HbA1c <10.1%).
* Stable concomitant medications defined as no changes in regimen for at least 2 weeks prior to Period 1 (daily adjustments of insulin doses are permitted).
* Body mass index of 18-40 kg/m².

Key Exclusion Criteria:

* Unable or unwilling to provide informed consent or to comply with study procedures.
* History of gastric surgery such as fundoplication, gastrectomy, gastric pacemaker placement, vagotomy, bariatric procedure. (Note: history of diagnostic endoscopy is not exclusionary).
* Acute or chronic illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the patient or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, poor renal or hepatic function, etc.
* Any clinically significant abnormalities on screening laboratories as determined by the Investigator.
* Abnormal 12-lead electrocardiogram (ECG), including evidence of acute myocardial or subendocardial ischemia and clinically significant arrhythmias or conduction abnormalities or blood pressure at screening except minor deviations deemed to be of no clinical significance by the Investigator.
* Poor venous access or inability to tolerate venipuncture.
* Acute GI illness within 48 hours of Period 1.
* Positive pregnancy test.
* Participation in a clinical study within the 30 days prior to dosing in the present study.
* Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic (PD) effects of RM-131 on gastric emptying | Day 1 at baseline vs Day 1 at 6 hours after dosing in Period 1 and Day 1 at baseline vs Day 1 at 6 hours after dosing in Period 2
  Change from baseline in gastric half-emptying time by scintigraphy (solids and liquids)

SECONDARY OUTCOMES:
Safety and tolerability of RM-131 | Day 1 and 2 after dosing in Period 1 and Day 1 and 2 after dosing in Period 2
  Number of participants with adverse events
Pharmacokinetics (PK) of RM-131 | Day 1 at baseline vs Day 1 at 6 hours after dosing in Period 1 and Day 1 at baseline vs Day 1 at 6 hours after dosing in Period 2
  Median T-max of RM-131 levels in patients with type 2 diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Shin A, Camilleri M, Busciglio I, Burton D, Smith SA, Vella A, Ryks M, Rhoten D, Zinsmeister AR. The ghrelin agonist RM-131 accelerates gastric emptying of solids and reduces symptoms in patients with type 1 diabetes mellitus. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1453-1459.e4. doi: 10.1016/j.cgh.2013.04.019. Epub 2013 Apr 30. PMID 23639598
- [Derived] Shin A, Camilleri M, Busciglio I, Burton D, Stoner E, Noonan P, Gottesdiener K, Smith SA, Vella A, Zinsmeister AR. Randomized controlled phase Ib study of ghrelin agonist, RM-131, in type 2 diabetic women with delayed gastric emptying: pharmacokinetics and pharmacodynamics. Diabetes Care. 2013 Jan;36(1):41-8. doi: 10.2337/dc12-1128. Epub 2012 Sep 6. PMID 22961573